CLINICAL TRIAL: NCT01896856
Title: A Phase I Study of SGI-110 Combined With Irinotecan Followed by a Randomized Phase II Study of SGI-110 Combined With Irinotecan Versus Regorafenib or TAS-102 in Previously Treated Metastatic Colorectal Cancer Patients
Brief Title: Phase I/II Study of SGI-110 With Irinotecan Versus Regorafenib or TAS-102 in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Van Andel Research Institute (Other); Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1369; NA_00085870 (Other: JHMIRB)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-08

CONDITIONS: Previously Treated Metastatic Colorectal Cancer
Keywords: SGI-110; irinotecan; regorafenib; methylation; colorectal; metastatic; TAS-102; lonsurf
MeSH Terms: conditions — Neoplasm Metastasis | interventions — guadecitabine; regorafenib; trifluridine tipiracil drug combination; Irinotecan

STUDY DESIGN:
Intervention Model Description: In Phase 2, Arm B patients who have disease progression will be given the option to receive Arm A study drugs.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1: Dose Escalation (Experimental): Subjects receive SGI-110 on days 1-5 and irinotecan on days 8 and 15 of each 28-day cycle.
  Various doses of SGI-110 are tested to determine the maximum tolerated dose in combination with irinotecan.
  Interventions: Drug: SGI-110 Dose Escalation
- Phase 2: Arm A SGI-110 + irinotecan (Experimental): Subjects receive SGI-110 on days 1-5 and irinotecan on days 8 and 15 of each 28-day cycle.
  Growth factor support (filgrastim and peg-filgrastim) is given during cycle 1 with option to give additional growth factor support at subsequent cycles per clinician judgement.
  Interventions: Drug: SGI-110; Drug: Irinotecan
- Phase 2: Arm B regorafenib or TAS-102 (Active Comparator): Subjects received either regorafenib or TAS-102 based on physician and patient preference. Subjects that had received one of these standard of care drugs (regorafenib or TAS-102) prior to enrollment received the other on study.
  Regorafenib taken daily from days 1-21 of each 28-day cycle or TAS-102 taken twice daily on days 1-5 and 8-12 of each 28-day cycle.
  Subjects who had disease progression on Arm B were given the option to receive Arm A study drugs after a 14 day wash-out period.
  Interventions: Drug: Regorafenib; Drug: TAS-102; Drug: SGI-110; Drug: Irinotecan

INTERVENTIONS:
Drug: SGI-110 Dose Escalation — * Dose level 1 (DL1): 45 mg/m^2 administered as a subcutaneous injection
  * Dose level 1G (DL1G): 45 mg/m^2 administered as a subcutaneous injection + growth factor support
  * Dose level -1 (DL-1): 30 mg/m^2 administered as a subcutaneous injection
  * Dose level -1G (DL-1G): 30 mg/m^2 administered as a subcutaneous injection + growth factor support
  Other Names: Guadecitabine
  Arms: Phase 1: Dose Escalation
Drug: Regorafenib — 160 mg taken orally
  Other Names: Stivarga
  Arms: Phase 2: Arm B regorafenib or TAS-102
Drug: TAS-102 — 35 mg/m^2 taken orally
  Other Names: Lonsurf; trifluridine and tipiracil
  Arms: Phase 2: Arm B regorafenib or TAS-102
Drug: SGI-110 — 45 mg/m^2 administered as a subcutaneous injection
  Other Names: Guadecitabine
  Arms: Phase 2: Arm A SGI-110 + irinotecan; Phase 2: Arm B regorafenib or TAS-102
Drug: Irinotecan — 125 mg/m^2 administered IV
  Other Names: Camptosar
  Arms: Phase 2: Arm A SGI-110 + irinotecan; Phase 2: Arm B regorafenib or TAS-102

SUMMARY:
This is a phase I/II study of the combination of Guadecitabine (SGI-110) and previously treated metastatic colorectal cancer patients. This study will be conducted in two components. First, patients will be enrolled in a phase I study of SGI-110 combined with irinotecan in a standard 3+3 design. After the maximum tolerated dose (MTD) is determined, patients will subsequently be enrolled in a 2:1 randomized phase II study of SGI-110 and irinotecan versus the standard of care regorafenib or Lonsurf (TAS-102).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum
* Phase I only: patients with biopsiable disease amenable to having two research biopsies.
* Have measurable disease
* Phase II only: progressed while receiving irinotecan therapy in the metastatic setting. There are no limitations on number of prior therapies in the metastatic setting.
* Life expectancy of greater than 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status <1
* Normal organ and marrow function as defined by study-specified laboratory tests
* Must use adequate contraception through the study and for 3 months after last dose of study drug.

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) of first dose of study drug or who have not recovered from treatment-related adverse events
* Receiving any other investigational agents
* Participants with known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to irinotecan, decitabine or SGI-110.
* Received prior therapy with any hypomethylating agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing women
* History of a different malignancy are ineligible with exceptions (disease-free for at least 5 years with low risk for recurrence, cervical cancer in situ, definitively treated early stage prostate cancer, definitively treated breast ductal or lobular carcinoma in situ, and basal cell or squamous cell carcinoma of the skin).
* HIV-positive individuals on combination antiretroviral therapy
* Phase II only: previous treatment with regorafenib and TAS-102. If patients have previously received either regorafenib OR TAS-102, they must be able to receive the alternate regimen if randomized to standard of care (Arm B).
* Hospitalization for an acute medical issue within 4 weeks prior to screening visit
* Symptomatic bowel obstruction within 6 months prior to enrollment, Patients who undergo surgical correction of obstructing lesion will be eligible within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-10-23 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilo Azad, MD, Principal Investigator — SKCCC at JHMI
Locations (4):
- United States (3):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
- VU Medisch Centrum, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee V, Parkinson R, Zahurak M, Cope L, Cercek A, Verheul H, Gootjes E, Lenz HJ, Iqbal S, Jones P, Baylin S, Rami V, Ahuja N, El Khoueiry A, Azad NS. A phase II study of guadecitabine combined with irinotecan vs regorafenib or TAS-102 in irinotecan-refractory metastatic colorectal cancer patients. Int J Cancer. 2024 May 15;154(10):1794-1801. doi: 10.1002/ijc.34845. Epub 2024 Feb 5. PMID 38312102
- [Derived] Sharma A, Vatapalli R, Abdelfatah E, Wyatt McMahon K, Kerner Z, A Guzzetta A, Singh J, Zahnow C, B Baylin S, Yerram S, Hu Y, Azad N, Ahuja N. Hypomethylating agents synergize with irinotecan to improve response to chemotherapy in colorectal cancer cells. PLoS One. 2017 Apr 26;12(4):e0176139. doi: 10.1371/journal.pone.0176139. eCollection 2017. PMID 28445481

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Dose Level 1: Guadecitabine (SGI-110) 45 mg/m^2 was administered as a subcutaneous injection on days 1-5 of each 28-day cycle. Irinotecan 125 mg/m^2 was administered IV on days 8 and 15 of each 28-day cycle.
- Phase 1: Dose Level -1: Guadecitabine (SGI-110) 30 mg/m^2 was administered as a subcutaneous injection on days 1-5 of each 28-day cycle. Irinotecan 125 mg/m^2 was administered IV on days 8 and 15 of each 28-day cycle.
- Phase 1: Dose Level -1G: Guadecitabine (SGI-110) 30 mg/m^2 was administered as a subcutaneous injection on days 1-5 of each 28-day cycle. Irinotecan 125 mg/m^2 was administered IV on days 8 and 15 of each 28-day cycle.
  Growth factor support (filgrastim and peg-filgrastim) mandatory during cycle 1, and given per clinician judgement cycle 2 and beyond.
- Phase 1: Dose Level 1G: Guadecitabine (SGI-110) 45 mg/m^2 was administered as a subcutaneous injection on days 1-5 of each 28-day cycle. Irinotecan 125 mg/m^2 was administered IV on days 8 and 15 of each 28-day cycle.
  Growth factor support (filgrastim and peg-filgrastim) mandatory during cycle 1, and given per clinician judgement cycle 2 and beyond.
- Phase 2: Arm A SGI-110 + Irinotecan: SGI-110 45 mg/m^2 was administered as a subcutaneous injection on days 1-5 of each 28-day cycle. Irinotecan 125 mg/m^2 was administered IV on days 8 and 15 of each 28-day cycle. Growth factor support (filgrastim and peg-filgrastim) was given during cycle 1 with option to give additional growth factor support at subsequent cycles per clinician judgement.
- Phase 2: Arm B Regorafenib or TAS-102: Subjects received either regorafenib or Lonsurf (TAS-102). Regorafenib 160 mg was taken orally daily from days 1-21 of each 28-day cycle or TAS-102 35 mg/m^2 was taken orally twice daily on days 1-5 and 8-12 of each 28-day cycle.
  Subjects that had previously received one of these standard of care drugs (regorafenib or TAS-102) received the other on study. For subjects that had never received either regorafenib or TAS-102, the choice of therapy was deferred to the treating physician and patient.
Period: Overall Study
Arm/Group | Phase 1: Dose Level 1 | Phase 1: Dose Level -1 | Phase 1: Dose Level -1G | Phase 1: Dose Level 1G | Phase 2: Arm A SGI-110 + Irinotecan | Phase 2: Arm B Regorafenib or TAS-102
Started | 6 | 3 | 7 | 6 | 62 | 34
Completed | 6 | 3 | 6 | 6 | 62 | 34
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Transportation issues / Non-compliance | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 2: Arm B Regorafenib or TAS-102: Subjects received either regorafenib or TAS-102. Regorafenib 160 mg was taken orally daily from days 1-21 of each 28-day cycle or TAS-102 35 mg/m^2 was taken orally twice daily on days 1-5 and 8-12 of each 28-day cycle.
  Subjects that had previously received one of these standard of care drugs (regorafenib or TAS-102) received the other on study. For subjects that had never received either regorafenib or TAS-102, the choice of therapy was deferred to the treating physician and patient.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Dose Level 1 | Phase 1: Dose Level -1 | Phase 1: Dose Level -1G | Phase 1: Dose Level 1G | Phase 2: Arm A SGI-110 + Irinotecan | Phase 2: Arm B Regorafenib or TAS-102 | Total
Number analyzed (Participants) | 6 | 3 | 7 | 6 | 62 | 34 | 118
Age, Continuous [Median (Full Range); unit: years] | 54.5 [47 to 69] | 64 [63 to 74] | 52 [41 to 72] | 54.5 [39 to 74] | 55.0 [29 to 80] | 59.5 [31 to 78] | 57.0 [29 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 4 | 21 | 18 | 49
  Male | 4 | 1 | 5 | 2 | 41 | 16 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 5 | 1 | 6
  Not Hispanic or Latino | 6 | 3 | 7 | 6 | 57 | 33 | 112
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 9 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 5 | 0 | 3 | 8 | 16
  White | 6 | 3 | 2 | 5 | 47 | 22 | 85
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Dose Limiting Toxicity
Description: Number of participants experiencing a Dose Limiting Toxicity (DLT) in each dose level. DLT is defined as any of the following study drug-related toxicities occurring during the first cycle of study drug on study:
  1. grade 4 thrombocytopenia lasting >7days
  2. any grade 3-4 febrile neutropenia
  3. grade 3 or higher non-hematologic toxicity unless it could be managed by supportive treatment
  4. any other clinically significant adverse event which would place subjects at undue safety risk, or results in discontinuation of treatment.
Time Frame: 28 days
Population: Per protocol, Dose Limiting Toxicities were only assessed in Phase 1 subjects in order to determine the Phase 2 dose of SGI-110. 1 Patient in Dose Level -1G was taken off study for non-compliance due to transportation issues before completion of Cycle 1 and was not considered evaluable for DLT analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: SGI-110 45 mg/m^2 subcutaneously on days 1-5 of each 28-day cycle Irinotecan 125 mg/m^2 IV on days 8 and 15 of each 28-day cycle.
- Dose Level -1: SGI-110 30 mg/m^2 subcutaneously on days 1-5 of each 28-day cycle Irinotecan 125 mg/m^2 IV on days 8 and 15 of each 28-day cycle.
- Dose Level -1G: SGI-110 30 mg/m^2 subcutaneously on days 1-5 of each 28-day cycle Irinotecan 125 mg/m^2 IV on days 8 and 15 of each 28-day cycle. Growth Factor Support with Filgrastim and/or Pegfilgrastim given during Cycle 1 and in subsequent cycles per clinician judgement.
- Dose Level 1G: SGI-110 45 mg/m^2 subcutaneously on days 1-5 of each 28-day cycle Irinotecan 125 mg/m^2 IV on days 8 and 15 of each 28-day cycle. Growth Factor Support with Filgrastim and/or Pegfilgrastim given during Cycle 1 and in subsequent cycles per clinician judgement.
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -1G | Dose Level 1G
Number analyzed (Participants) | 6 | 3 | 6 | 6
Participants | 1 | 2 | 1 | 1

2. Primary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival is the time (in months) from start of treatment to progression, clinical deterioration attributed to disease, or death.
Time Frame: Up to 12 months
Population: Per protocol, the progression-free survival objective was only assessed in Phase 2 subjects. 18 subjects who received Arm B treatment were eligible to "crossover" to receive Arm A treatment. These participants were not included in the number analyzed in Arm A because they were not assessed for progression free survival after Arm A treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Arm A SGI-110 + Irinotecan | Phase 2: Arm B Regorafenib or TAS-102
Number analyzed (Participants) | 62 | 34
months | 2.37 [2.2 to 3.52] | 2.09 [1.91 to 2.99]

3. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time (in months) between the start of treatment and death.
Time Frame: Up to 3 years
Population: Per protocol, the overall survival objective was only assessed in Phase 2 subjects. 18 subjects who received Arm B treatment and were eligible to "crossover" to receive Arm A treatment were not included in the number analyzed in Arm A because they were not assessed for overall survival after receiving Arm A treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Arm A SGI-110 + Irinotecan | Phase 2: Arm B Regorafenib or TAS-102
Number analyzed (Participants) | 62 | 34
months | 7.15 [6.6 to 8.02] | 7.66 [4.83 to 9.36]

4. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate (ORR) is defined as the number of subjects achieving a Complete Response (CR) or Partial Response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. CR = disappearance of all target lesions, PR = at least 30% decrease in the sum of diameters of target lesions.
Time Frame: Assessed until disease progression, up to 3 years
Population: ORR only assessed for Phase 2. 5 from Arm A and 2 from Arm B were excluded from response rate analysis as they didn't get a follow-up scan. 18 subjects in Arm B were eligible to "crossover" to receive Arm A treatment. They were not included in the number analyzed in Arm A because they were not assessed for objective response after Arm A treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Arm A SGI-110 + Irinotecan | Phase 2: Arm B Regorafenib or TAS-102
Number analyzed (Participants) | 57 | 32
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the first dose of study drug through 30 days after the last dose of study drug, up to 13 months
Description: 18 patients from Arm B were eligible to "crossover" to receive Arm A study treatment after they had progression with Arm B treatment. They were assessed for adverse events after receiving Arm A treatment. Their adverse events are reported here in a separate arm.
Groups:
- Phase 2: "Crossover" to Arm A From Arm B: Per protocol, Arm B subjects were given the option to "crossover" and receive Arm A study drugs after disease progression on Arm B.
  18 Arm B subjects received Arm A study drugs after initial progression.
  SGI-110 45 mg/m^2 was administered as a subcutaneous injection on days 1-5 of each 28-day cycle. Irinotecan 125 mg/m^2 was administered IV on days 8 and 15 of each 28-day cycle. Growth factor support (filgrastim and peg-filgrastim) was given during cycle 1 with option to give additional growth factor support at subsequent cycles per clinician judgement.
Arm/Group | Phase 1: Dose Level 1 | Phase 1: Dose Level -1 | Phase 1: Dose Level -1G | Phase 1: Dose Level 1G | Phase 2: Arm A SGI-110 + Irinotecan | Phase 2: "Crossover" to Arm A From Arm B | Phase 2: Arm B Regorafenib or TAS-102
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/7 | 1/6 | 3/62 | 0/18 | 4/34
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/3 | 2/7 | 1/6 | 15/62 | 8/18 | 1/34
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 6/7 | 6/6 | 58/62 | 18/18 | 30/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Dose Level 1 (N=6) | Phase 1: Dose Level -1 (N=3) | Phase 1: Dose Level -1G (N=7) | Phase 1: Dose Level 1G (N=6) | Phase 2: Arm A SGI-110 + Irinotecan (N=62) | Phase 2: "Crossover" to Arm A From Arm B (N=18) | Phase 2: Arm B Regorafenib or TAS-102 (N=34)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 4 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue or Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Fever (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 3 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Dose Level 1 (N=6) | Phase 1: Dose Level -1 (N=3) | Phase 1: Dose Level -1G (N=7) | Phase 1: Dose Level 1G (N=6) | Phase 2: Arm A SGI-110 + Irinotecan (N=62) | Phase 2: "Crossover" to Arm A From Arm B (N=18) | Phase 2: Arm B Regorafenib or TAS-102 (N=34)
Anemia (Blood and lymphatic system disorders) | 4 | 2 | 5 | 2 | 37 | 8 | 15
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 5 | 1 | 4 | 3 | 7 | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 6 | 3 | 5 | 4 | 27 | 10 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 3 | 2 | 20 | 6 | 3
Leukopenia (Blood and lymphatic system disorders) | 6 | 1 | 5 | 4 | 28 | 6 | 11
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Glucose intolerance (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 5 | 3 | 6
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 4 | 1 | 3
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 3 | 3 | 24 | 6 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 6 | 4 | 28 | 5 | 11
Vomiting (Gastrointestinal disorders) | 0 | 3 | 4 | 2 | 9 | 4 | 5
Chills (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 1 | 0 | 4 | 1 | 1 | 0 | 0
Fatigue or malaise (General disorders) | 3 | 2 | 4 | 5 | 37 | 10 | 14
Fever (General disorders) | 4 | 1 | 2 | 0 | 8 | 0 | 1
Injection site reaction (General disorders) | 4 | 1 | 5 | 4 | 12 | 5 | 0
Abscess or skin infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 3 | 1 | 5 | 2 | 8 | 0 | 0
ALT increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 3
AST increased (Investigations) | 2 | 0 | 4 | 1 | 2 | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 5 | 1 | 2
Weight loss (Investigations) | 1 | 0 | 0 | 0 | 5 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 0 | 3 | 3 | 14 | 2 | 11
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1
Hyperglycemia (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Hypocalcemia (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypophosphatemia (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 3 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 0 | 3 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 1 | 0 | 3 | 0 | 2
Headache (Nervous system disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 2 | 11 | 1 | 1
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigators (PIs) from participating sites must provide the Johns Hopkins PI with a copy of any proposed publication for review and comment at least 30 days prior to submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT01896856/Prot_SAP_000.pdf